CLINICAL TRIAL: NCT07341321
Title: SARS-CoV-2 mRNA Vaccination in Patients With Hepatocellular Carcinoma Treated With Immune Checkpoint Inhibitors (CoVaCheck) A Multicenter Retrospective Cohort Analysis in Austria
Brief Title: SARS-CoV-2 mRNA Vaccination in Patients With Hepatocellular Carcinoma Treated With Immune Checkpoint Inhibitors
Acronym: CoVaCheck
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Klinikum Wels-Grieskirchen (Other); University Hospital St. Polten (Other); Ordensklinikum Linz GmbH Krankenhaus Barmherzige Schwestern (Unknown); Krankenhaus der Barmherzigen Brüder St. Veit/Glan (Unknown)
Responsible Party: Sponsor
Other Study IDs: CoVaCheck
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: mRNA Vaccination; Hepatocellular Carcinoma; Checkpoint Inhibitor
Keywords: hepatocellular carcinoma; mRNA vaccination; response; immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccinated: Patients with hepatocellular carcinoma, undergoing checkpoint inhibitor therapy, vaccinated with mRNA vaccine within last 100 days
- not vaccinated: Patients with hepatocellular carcinoma, undergoing checkpoint inhibitor therapy, not vaccinated with mRNA vaccine within last 100 days

SUMMARY:
A multicenter retrospective cohort analysis in Austria

Primary Objective:

To assess whether receiving an mRNA COVID-19 vaccine within 3 months before starting ICI (Immune checkpoint inhibitors) therapy improves best overall response (mRECIST) in HCC (hepatocellular carcinoma).

Secondary Objectives:

Evaluate whether vaccination within 1 or 3 months affects OS (overall survival) , PFS (Progression free survival)), or TTP (Time to progression); compare outcomes by vaccination status, vaccine type, and prior infection; explore modification by cirrhosis severity and tumor characteristics; and assess safety (irAEs, steroid use, toxicity-related discontinuation).

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) have become a cornerstone of systemic therapy for advanced hepatocellular carcinoma (HCC). Their efficacy, however, varies substantially between patients, and factors that modulate immunotherapy response remain incompletely understood .

Recent mechanistic and clinical data have raised the hypothesis that SARS-CoV-2 mRNA vaccines might augment responsiveness to ICIs. A landmark study by Grippin et al. demonstrated that mRNA vaccines induce a systemic surge of type-I interferons, activate antigen-presenting cells, increase PD-L1 expression on tumor cells, and ultimately sensitize tumors to ICIs across various malignancies including NSCLC (non-small cell lung cancer) and melanoma. In their retrospective cohorts, receiving a COVID-19 mRNA vaccine within 100 days before starting ICI was associated with significantly improved overall survival and progression-free survival While these findings suggest that COVID-19 mRNA vaccines may act as potent immune modulators in the context of immunotherapy, no data exist for HCC, a tumor entity that is characterized by an immunosuppressive, 'immune-cold' microenvironment that limits effective anti-tumor immune responses.

Given the widespread implementation of COVID-19 vaccination programs in Austria since 2021, and the large number of HCC patients receiving ICI-based therapies at tertiary centers, a rigorous retrospective analysis is now feasible.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Radiologically or histologically confirmed hepatocellular carcinoma
* Treatment with immune checkpoint inhibitor-based therapy (mono- or combination therapy; e.g., atezolizumab/bevacizumab, durvalumab/tremelimumab, nivolumab, pembrolizumab)
* Complete electronic medical records available
* At least one imaging-based response assessment using mRECIST

Exclusion Criteria:

* Missing key clinical data required for main analyses (e.g. survival status, date of progression, Child-Pugh class, BCLC stage)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all eligible patients with HCC treated within the past 5 years (January 2021 - December 2025, depending on center availability) with one of the specified checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Best overall response | up to 4 years
  according to mRECIST criteria

SECONDARY OUTCOMES:
Overall survival | up to 4 years
  death yes/no
Progression free survival | up to 4 years
  Progression according to RECIST yes/no
Time to progression | up to 4 years
  Time until progression occurs according to RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Florian Rainer, MD, Principal Investigator — Medizinische Universität Graz; Vanessa Stadlbauer, Univ Prof, Principal Investigator — Medizinische Universität Graz; Walter Spindelböck, MD, Principal Investigator — Medizinische Universität Graz
Locations (5):
- Austria (5):
  - Medical University of Graz, Graz
  - Ordensklinikum Linz, Linz
  - University Hospital St. Pölten, Sankt Pölten
  - Krankenhaus der Barmherzigen Brüder St Veit an der Glan, Sankt Veit an der Glan
  - Klinikum Wels-Grieskirchen, Wels

IPD SHARING:
Plan to Share IPD: Yes
Upon request and after having a data sharing agreement in place, pseudonymized IPD can be shared.